CLINICAL TRIAL: NCT06572839
Title: A Randomized Controlled Multicenter Trial, Examining the Effect of Amnio-Maxx on the Healing Rate of Chronic Diabetic Foot Ulcers
Brief Title: Amnio-Maxx in Patients With Diabetic Foot Ulcers Unresponsive to Standard of Care Treatment Alone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capsicure, LLC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Med-Maxx
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Foot Ulcer
Keywords: chronic ulcers; wound care; Dual Layer Amnion Patch
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: The patient will be randomized to standard of care (SOC) or Amnio-Maxx as an addition to SOC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No intervention: Standard of Care (No Intervention): Debridement, offloading, and proper moisture balance dressings
- Amnio-Maxx as an addition to standard of care (Experimental): Device exposure is estimated to be a maximum of 12 weeks
  Interventions: Other: Amnio-Maxx

INTERVENTIONS:
Other: Amnio-Maxx — Amnio-Maxx Dual Layer Amnion Patch is processed using aseptic techniques, treated with a saline solution and dehydrated.
  Other Names: Amnio-Maxx Dual Layer Amnion Allograft
  Arms: Amnio-Maxx as an addition to standard of care

SUMMARY:
This randomized controlled study evaluates the adjuvant use of Amnio-Maxx in patients with diabetic foot ulcers

DETAILED DESCRIPTION:
This is a multicenter randomized open-label clinical study in patients with Wagner grade 1 and 2 DFUs. Diabetic patients presenting with chronic nonhealing ulcers will be screened for eligibility. At least 50% of the eligible population will be drawn from patients ≥ 65 years of age. All patients will complete a 2-week run-in period prior to treatment allocation to Amnio-Maxx and standard of care (SOC) or SOC alone. Patients will be seen at weekly intervals (± 3 days) for the 12 weeks treatment period. If additional dressing changes are required between the scheduled visits, the occurrence of these visits will be recorded. Primary efficacy endpoints include percentage change in ulcer size at 12 weeks along with the proportion of participants achieving complete wound closure. Additionally, pain and safety will be assessed as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are 18 years of age or older. At least 50% of the enrolled population must be > 65 years of age.
2. Subject history of Type I or Type II Diabetes Mellitus requiring oral glycemic control and/or insulin replacement therapy.
3. Subjects with the following ulcer:

   A. Presence of a DFU Wagner 1 or 2 grade at the first screening visit on any aspect of the foot, provided it is at or below the aspect of the medial malleolus. [NOTE: If two or more DFUs are present with the same grade, the index ulcer is the largest ulcer and the only one evaluated in the study. Index ulcer must be more than 5 cm distant apart.

   B. A DFU is present for greater than 4 weeks (documented in the medical record) but less than 12 months duration if being treated with active SOC.
4. Objectively, less than 20% healing in the two-week screening period prior to randomization.
5. Study ulcer is a minimum of 1.0 cm2 and a maximum of 25 cm2 post-debridement at first treatment visit
6. Index ulcer and/or index ulcer limb may have had prior infection, but infection(s) must be adequately treated and controlled as defined by IDSA Guidelines Grade level 1.
7. The subject is able and willing to follow the protocol requirements.
8. Subject has signed informed consent.
9. Adequate circulation to the affected foot as demonstrated by a dorsum transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg; an ABI between 0.7 and ≤ 1.3, or TBI of >6 within 3 months of the first Screening Visit.
10. Negative pregnancy test for females of childbearing potential (e.g., not post- menopausal for at least one year or surgically sterile). Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence) starting at Screening and continuing through the duration of their study participation.
11. The index ulcer has been offloaded with protocol defined offloading device throughout the study run-in period for at least 14 days prior to randomization (Run- in period defined as Screening through TV1/Randomization).
12. The index ulcer has a clean base and free of necrotic debris at time of placement of treatment product.

Exclusion Criteria:

1. Subject has a documented life expectancy of < 1 year.
2. Index ulcer has been present for >1 year.
3. Patient does not have adequate 2-week historical data demonstrating < 20% area reduction.
4. Subject is unable to comply with offloading device.
5. Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence to medical treatment.
6. Subject has ulcers that are completely necrotic or fibrotic tissue.
7. Subject has major uncontrolled medical disorders such as serious cardiovascular, renal, liver or pulmonary disease, lupus, palliative care or sickle cell anemia.
8. Subject currently being treated for an active malignant disease or subjects with history of malignancy within the ulcer.
9. The Subject has other concurrent conditions that in the opinion of the Principal Investigator may compromise subject safety.
10. Known contraindications to amniotic tissue membranes or known allergies to any of the Amnio-Maxx components.
11. Concurrent participation in another clinical trial that involves an investigational drug or device that would interfere with this study.
12. Index ulcer has reduced in area by 20% or more after 2 weeks of SOC from the first screening visit (S1) to the TV1/randomization visit.
13. Subject is pregnant or breastfeeding.
14. Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within 30 days prior to randomization visit or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
15. Index ulcer has been previously treated with tissue engineered materials (e.g. Apligraf® or Dermagraft®) or other scaffold materials (e.g. Oasis, Matristem) within the last 30 days preceding the first treatment visit.
16. Affected extremity requiring hyperbaric oxygen during the trial or within 2 weeks of screening treatment visit 1.
17. Presence of diabetes with poor metabolic control as documented with an HbA1c ≥12.0 within 30 days of randomization (TV1).
18. Index ulcer and/or index limb with presence of, gangrene or unstable ischemia at screening (SV1).
19. Revascularization surgery on the lower extremity on which the index ulcer is located within 30 days of Screening Visit (SV1).
20. Index ulcer in the opinion of the Principal Investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a neoplasm of the ulcer.
21. Any clinically significant finding, in the judgment of the Principal Investigator, that would place the subject at health risk, impact the study, or affect the completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Wound Closure Assessment Verified with Independent Adjudication | 12 weeks
  To demonstrate change in healing rates of chronic wounds (diabetic foot ulcers), unresponsive to standard therapy.
Percentage Area Reduction verified with Independent Adjudication | 12 weeks
  To demonstrate change in healing rates of chronic wounds (diabetic foot ulcers), unresponsive to standard therapy.

SECONDARY OUTCOMES:
Chage of Subjects Pain Levels | 12 weeks
  Subject pain assessed through the Numeric Pain Rating Scale on a weekly basis throughout the study
Change in Adverse Events | 12 weeks
  Change in Adverse Events estimated from the observed data through physician reporting

CONTACTS AND LOCATIONS:
Overall Officials: Windy Cole, DPM, Principal Investigator — Capsicure, LLC; Marissa Docter, RN, BSN, MD, Study Director — Capsicure, LLC
Locations (12):
- United States (12):
  - North Alabama Research Center, LLC, Athens, Alabama
  - North Park Podiatry, San Diego, California
  - Solutions Medical Research, Coral Gables, Florida
  - Evolution Research Center, Hialeah, Florida
  - Symphony Research, Jacksonville, Florida
  - Quality Care Clinical Research, Miami, Florida
  - Medcentris, Hammond, Louisiana
  - Curalta Clinical Trials, Oradell, New Jersey
  - Suffolk Foot and Ankle, East Patchogue, New York
  - PA Foot and Ankle Associates, Allentown, Pennsylvania
  - Stride Clinical Research, Houston, Texas
  - Ten20 Medical, Sunnyvale, Texas

IPD SHARING:
Plan to Share IPD: No
Neither the complete nor any part of the results of the study carried out under this protocol, nor any of the information provided by the sponsor for the purposes of performing the study, will be published or passed on to any third party without the consent of the study sponsor. Any investigator involved with this study is obligated to provide the sponsor with complete test results and all data derived from the study.